CLINICAL TRIAL: NCT03752814
Title: SYNOSTE Nitinail System Trial
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study was stopped due to administrative reasons.
Sponsor: SYNOSTE Oy (Industry)
Collaborators: MVZ Labor Dr. Limbach (Unknown); Technical University of Munich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-2017
Record Dates: First submitted 2018-11-16; First posted 2018-11-26 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Leg Length Inequality
Keywords: distraction osteogenesis; bone lengthening; leg length discrepancy; callotasis; Intramedullary distraction nail
MeSH Terms: conditions — Leg Length Inequality

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYNOSTE Nitinail System (Experimental): The intended purpose of the SNS in this trial is lengthening of the femur by callotasis.
  Interventions: Device: SYNOSTE Nitinail System

INTERVENTIONS:
Device: SYNOSTE Nitinail System — Mode of application: 1. Implantation surgery: osteotomy and antegrade implantation of SNS in femur for distraction osteogenesis (callotasis), 2. distraction osteogenesis (implant lengthening phase), 3. Bone healing (implant as stabilizing element during consolidation phase), 4. Explantation after consolidation.

SUMMARY:
SYNOSTE Nitinail System Trial is an international multicenter open label single-arm equivalence study to verify whether the leg-lengthening procedure can be adequately controlled with the SNS system as measured with the lengthening control index (LCI) at the end of the distraction period.

DETAILED DESCRIPTION:
The SYNOSTE Nitinail System (SNS) is an assembly of an active implantable distraction nail (SYNOSTE Nitinail), Locking screws, accessory instruments for surgery and the home care unit (also External control unit (ECU) or Halo). It includes also, a software tool, Syndex, that supports setting up the number of lengthening activations needed per day.

The SNS is intended for lengthening of the femur by distraction osteogenesis.

The study will consist of a recruitment period of 3 months and an observation period of roughly 24 months (6 months after explantation). The observation period is split in two parts: The first part contains the most critical treatment phases from implantation surgery of the device through the actual lengthening phase up to the end of the bone healing. The second part contains only two visits: the explantation surgery of the device and a control at 6 months of further follow-up.

After the fist part of the trial, a primary analysis of the data including the hypothesis testing will be carried out. After the second part of the trial a follow-up analysis will be done.

16 (max 20) patients will be recruited in Finland and Turkey.

ELIGIBILITY:
Inclusion Criteria:

* Indication for femoral lengthening from different etiologies of max. 70 mm at single lengthening
* 18 to 65 years regardless of gender
* Suitable anatomy for SNS
* Able and willing to comply with study procedures

Exclusion Criteria:

* Other electronic implants
* Other Metallic implants in the affected limb below the osteotomy level
* Need for Magnetic Resonance imaging during the study
* BMI>30kg/m2 or weight>100kg
* Smoker
* Known hypersensitivity to Co, Ni, Cr or Ti metals
* Known hypersensitivity to Poly-Ether-Ether-Ketone (PEEK) or Ultrahigh Molecular Weight Poly-Ethylene (UHMWPE)
* Open growth plates
* Malignancy or tumor in bone
* Osteitis or soft tissue infection
* Significant existing deficit in range of motion of the adjacent joints
* Pseudoarthrosis
* Pregnancy
* Low psychological compliance (e.g. drug abuse)
* Simultaneous bilateral lengthening
* Need for osteotomies at multiple levels

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Lengthening control index (LCI) | 2,5 months
  The primary objective is to verify whether the leg-lengthening procedure can be adequately controlled with the SNS system as measured with the lengthening control index (LCI) at the end of the distraction period defined as LCI = DIachieved / DIscheduled
  ,where DIachieved = Achieved distraction index, ie. the daily rate of distraction has on average occurred during the lengthening phase in mm/d. DIscheduled = mean scheduled lengthening rate in mm/day.
  Analyzed at primary analysis.

SECONDARY OUTCOMES:
Performance of Nitinail/Mechanical stability of Nitinail | 6-9 months
  Mechanical stability of Nitinail as defined by the ratio of the numbers of breakages (nail and screws) to total nails implanted (% and absolute values) at the end of consolidation
Performance of Nitinail/Nitinail lengthening target achieved (%) | 2,5 months
  Nitinail lengthening target achieved as defined by % of targeted lengthening achieved by Nitinail determined at the end of lengthening period
Performance of Nitinail/Nitinail lengthening target achieved (absolute value) | 2,5 months
  Nitinail lengthening target achieved as defined by absolute value of targeted lengthening achieved by Nitinail determined at the end of lengthening period
Performance of Nitinail/Translation of nail lengthening to bone lengthening (%) | 2,5 months
  Translation of nail lengthening to bone lengthening as % of the Bone gap increase from achieved lengthening of Nitinail determined at the end of lengthening period
Performance of Nitinail/Translation of nail lengthening to bone lengthening (absolute value) | 2,5 months
  Translation of nail lengthening to bone lengthening as absolute value of the Bone gap increase from achieved lengthening of Nitinail determined at the end of lengthening period
Performance of Nitinail/Retention of achieved length by Nitinail | 6-9 months
  Retention of achieved length by Nitinail as change of achieved lengthening of Nitinail between end of distraction and end of consolidation
Patient Reported Outcomes/Patient Satisfaction | 6-9 months AND 24 months
  Patient satisfaction as the overall satisfaction value from Numeric Rating Scale at end of consolidation and final follow-up. The NRS for overall outcomes is a undimensional measure of satisfaction intensity, where the patient selects among 0-10 integers to describe the intensity of their overall satisfaction with the treatment outcomes on a horizontal line. "0" represents completely dissatisfied and "10" fully satisfied
Patient Reported Outcomes/Patient Satisfaction (aesthetic outcomes) | 6-9 months AND 24 months
  Patient satisfaction as the aesthetic outcomes value from Numeric Rating Scale (NRS) at end of consolidation and final follow-up. The NRS for aesthetic outcomes is a undimensional measure of satisfaction intensity, where the patient selects among 0-10 integers to describe the intensity of their satisfaction with the aesthetic outcomes on a horizontal line. "0" represents completely dissatisfied and "10" fully satisfied.
Patient Reported Outcomes/Change in scores of 36-Item Short Form Survey (SF-36) | 6-9 months AND 24 months
  Change in scores of SF-36 from preoperative baseline to end of consolidation for Primary analysis and to last visit for the Follow-up analysis. The used version of the SF-36 is the RAND 36-item health survey 1.0 (1993) with a time frame of 4 weeks. The SF-36 is an established and widely used set of generic, coherent, and easily administered quality-of-life measures in adults. Scoring will be done according to the instructions provided by RAND. Single item scores as well as health concept scale scores range from 0 to 100. A higher score defines a more favorable health state, with a value of 100 representing full health.
Patient Reported Outcomes/Patient pain status | 2,5 months
  Patient pain status as change of Numeric Rating Scale (NRS) from preoperative baseline to End of distraction (2,5 months). The NRS for pain is a undimensional measure of pain intensity, where the patient selects among 0-10 integers to describe the intensity of their pain on a horizontal line. "0" represents no pain and "10" worst possible pain.
Patient Reported Outcomes/Patient pain status | 24 months
  Patient pain status as the pain profile of the Numeric Rating Scale (as described above) during the treatment (until 24 months)
Patient Reported Outcomes/Patient pain status (consumption of pain medication) | 24 months
  Patient pain status as consumption of pain medication
Patient Reported Outcomes/Length of sick leave due to treatment | 6-9 months AND 24 months
  Length of sick leave due treatment in days assessed until the end of consolidation and end of treatment for Primary and Follow-up analyses, respectively
Clinical Success of Treatment/Femur lengthening target achieved (%) | 6-9 months AND 24 months
  Femur lengthening target achieved as % of the achieved femoral length increase of the targeted femoral length increase in mm determined at the end of consolidation and end of treatment for Primary and Follow-up analyses
Clinical Success of Treatment/Femur lengthening target achieved (absolute value) | 6-9 months AND 24 months
  Femur lengthening target achieved as absolute value of the achieved femoral length increase of the targeted femoral length increase in mm determined at the end of consolidation and end of treatment for Primary and Follow-up analyses
Clinical Success of Treatment/Weight bearing index | 6-9 months
  Weight bearing index as time to final full weight bearing (in days) per the achieved femoral length increase (in cm)
Clinical Success of Treatment/Consolidation index | 6-9 months
  Consolidation index as time to radiological confirmation of 3 cortices bridging the bony gap (in days) per the achieved femoral length increase (in cm)
Clinical Success of Treatment/Knee and hip joint Range of Motion (ROM) | 6-9 months AND 24 months
  Knee and hip joint Range of Motion (ROM) as flexion and extension at preoperative baseline, End of distraction and End of consolidation and compared to normal population values
Nitinail System Safety/Number and type of device related (Serious)Adverse Events | (6-9 months AND 24 months)
  Number and type of device related (Serious)Adverse Events reported until the end of consolidation and end of treatment.
Nitinail System Safety/Duration of surgery | 10 days and 18 months
  Duration of surgery of Nitinail related surgeries from cut-to- closure in minutes
Nitinail System Safety/Length of hospital stay | 10 days and 18 months
  Length of hospital stay of Nitinail related surgeries in days the patient spent in hospital perioperatively.
Nitinail System Safety/Patient compliance to lengthening protocol | 2,5 months
  Patient compliance to lengthening protocol as ratio of lengthening periods with non- compliance to protocol with all lengthening periods with one patient.
Nitinail System Safety/Release of metallic ions from the Nitinail | 3 months/further monitoring up to 24 months
  Release of metallic ions from the Nitinail as Cobalt and Chromium ion concentrations in blood from preoperative baseline to end of distraction.

CONTACTS AND LOCATIONS:
Overall Officials: Metin Küçükkaya, Prof. Dr., Principal Investigator — Şişli Florence Nightingale Hospital, Şişli/İstanbul, Turkey; Jan Lindahl, Dr., Principal Investigator — HUCH Ortopedics and Traumatology, Töölö Hospital, Finland
Locations (2):
- HUCH Ortopedics and Traumatology, Töölö Hospital, Helsinki, Uusimaa, Finland
- Şişli Florence Nightingale Hospital, Şişli/İstanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No